CLINICAL TRIAL: NCT02535442
Title: An Exploratory Study to Evaluate the Microbial Consortia and the Host Inflammatory Factors Present in the Nasal Passages of Patients During Upper Respiratory Symptomology and When Healthy
Brief Title: Nasal Swab Study to Explore the Nasal Microbia
Status: Completed | Type: Observational
Sponsor: Kimberly-Clark Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 500-15-0003
Record Dates: First submitted 2015-08-14; First posted 2015-08-28 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: None Retained — microbiota from nasal samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to evaluate the microbial consortia and the host inflammatory factors present in the nasal passages of patients during upper respiratory symptomology and when healthy using culture and molecular analysis techniques.

ELIGIBILITY:
Inclusion Criteria:

* Adults, male or female, between the ages 18 - 60
* Exhibiting symptoms of an upper respiratory ailment, which may include runny or stuffy nose, sore throat, fever, headache, cough, malaise, or loss of appetite with no indication or intention to treat with excluded medications.

Exclusion Criteria:

* Use of antibiotics, antifungals, antivirals, antihistamines, anticholinergic, anti-inflammatory, any nasal inhaled medications (other than saline), or steroid medications within the four (4) weeks prior to enrollment and during the course of the study. Use of cough suppressants and herbal medications are permitted.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample of male and female subjects with common cold symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2015-08; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Type and amount of nasal microbes | Change from baseline compared to Day 21

CONTACTS AND LOCATIONS:
Overall Officials: Charles Fogarty, MD, Principal Investigator — Spartanburg Medical Research
Locations (1):
- Spartanburg Medical Research, Spartanburg, South Carolina, United States

REFERENCES:
- [Background] Wolcott RD, Dowd SE. A rapid molecular method for characterising bacterial bioburden in chronic wounds. J Wound Care. 2008 Dec;17(12):513-6. doi: 10.12968/jowc.2008.17.12.31769. PMID 19052515
- [Background] Dowd SE, Wolcott RD, Sun Y, McKeehan T, Smith E, Rhoads D. Polymicrobial nature of chronic diabetic foot ulcer biofilm infections determined using bacterial tag encoded FLX amplicon pyrosequencing (bTEFAP). PLoS One. 2008 Oct 3;3(10):e3326. doi: 10.1371/journal.pone.0003326. PMID 18833331
- [Background] Callaway TR, Dowd SE, Wolcott RD, Sun Y, McReynolds JL, Edrington TS, Byrd JA, Anderson RC, Krueger N, Nisbet DJ. Evaluation of the bacterial diversity in cecal contents of laying hens fed various molting diets by using bacterial tag-encoded FLX amplicon pyrosequencing. Poult Sci. 2009 Feb;88(2):298-302. doi: 10.3382/ps.2008-00222. PMID 19151343
- [Background] Wolcott RD, Gontcharova V, Sun Y, Dowd SE. Evaluation of the bacterial diversity among and within individual venous leg ulcers using bacterial tag-encoded FLX and titanium amplicon pyrosequencing and metagenomic approaches. BMC Microbiol. 2009 Oct 27;9:226. doi: 10.1186/1471-2180-9-226. PMID 19860898
- [Background] Dowd SE, Callaway TR, Wolcott RD, Sun Y, McKeehan T, Hagevoort RG, Edrington TS. Evaluation of the bacterial diversity in the feces of cattle using 16S rDNA bacterial tag-encoded FLX amplicon pyrosequencing (bTEFAP). BMC Microbiol. 2008 Jul 24;8:125. doi: 10.1186/1471-2180-8-125. PMID 18652685